CLINICAL TRIAL: NCT06977854
Title: A SINGLE CENTER, SINGLE-BLIND STUDY DESIGN IN HEALTHY SUBJECTS TO EVALUATE SEVERAL EFFECTS OF CITRULLINE SUPPLEMENTS
Brief Title: The Objective of This Study Was to Compare and Quantify the Bioavailability of Citrulline Byproducts in Blood Samples and in Urine Samples After a Single Dose of the Assigned Dietary Supplement. The Treatment Arms Containing the Following Molecules: Citrulline HCL and L-Citrulline,
Status: Completed | Type: Observational
Sponsor: Vireo Systems, Inc. (Industry)
Collaborators: Princeton Consumer Research (Other)
Responsible Party: Sponsor
Other Study IDs: VIRUSE2R
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Bioavailability and AUC
Keywords: Citrulline,Arginine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Generally healthy male and female subjects aged 18-64
  Interventions: Other: Removal from study. In case of adverse event, subject treated for the AE.; Other: removal from study

INTERVENTIONS:
Other: Removal from study. In case of adverse event, subject treated for the AE. — The participation of a subject in this study may have been discontinued for any of the following reasons:
  * the subject wished to withdraw from study participation;
  * if, in the opinion of the Investigator, it was in the best interest of the subject;
  * suspected adverse effects from the test article;
  * inter-current illness;
  * violation of the prohibitions and restrictions;
  * development of an exclusion criteria. Subjects were free to withdraw at any time and need not give a reason, however, every reasonable attempt was made to ascertain such reasons. The data for those subjects who were withdrawn was included in the final clinical report but may be excluded from final data analysis.
Other: removal from study — The participation of a subject in this study may have been discontinued for any of the following reasons:
  * the subject wished to withdraw from study participation;
  * if, in the opinion of the Investigator, it was in the best interest of the subject;
  * suspected adverse effects from the test article;
  * inter-current illness;
  * violation of the prohibitions and restrictions;
  * development of an exclusion criteria. Subjects were free to withdraw at any time and need not give a reason, however, every reasonable attempt was made to ascertain such reasons. The data for those subjects who were withdrawn was included in the final clinical report but may be excluded from final data analysis.

SUMMARY:
Citrulline dietary supplements are of interest for improving cardiovascular and exercise performance. The health benefits of citrulline are attributable to its ability to increase arginine levels in the body through the intestinal-renal arginine conversion pathway. From a dietary supplementation standpoint, citrulline offers advantages over arginine due to its reduced first-pass metabolism and ready conversion to arginine within the body. While L-citrulline is the most widely used citrulline dietary supplement, additional salt forms such as citrulline maleate and citrulline HCl may provide improvements in the delivery of arginine to the body. The present study compared the single-dose pharmacokinetics of L-citrulline and citrulline HCl formulations in healthy human subjects. A total of 17 subjects were randomly assigned to groups receiving either 6 g of L-citrulline, 6 g of citrulline HCl or 2 g of citrulline HCl. The resulting increases in citrulline and arginine in plasma and urine samples were determined using liquid chromatography-multiple reaction monitoring mass spectrometry (LC-MRM/MS). All citrulline dietary supplements examined produced time-dependent increases in plasma citrulline and arginine. Both maximal plasma concentration (Cmax) and area under the plasma vs time curve (AUC) for citrulline were modestly reduced in the 6 g citrulline HCl treatment group, the resulting arginine Cmax and AUCs were similar for both L-citrulline and citrulline HCl at the 6 g dose. While the 2 g dose of citrulline HCl had reduced Cmax and AUC values compared to 6 g doses, the time to reach peak levels of arginine were significantly shorter. Furthermore, examination of the relative arginine bioavailability achieved with the 6 g and 2 g citrulline HCl compared to the 6 g L-citrulline was approximately 120% and 215%, respectively, consistent with an improved citrulline to arginine conversion efficiency with the citrulline HCl formulations.

ELIGIBILITY:
Inclusion Criteria:

* healthy and hydrated male or female ages 18-64; agrees to refrain from citrulline-rich foods; able and willing to fast 12 hours prior to baseline visit; willing to have blood and urine collections as dictated in the protocol; females of child bearing age have some type of birth control.

Exclusion Criteria:

* female subject is pregnant; allergies or sensitivities to citrulline products; history of losing consciousness during blood collection;past medical history of iron deficiency; history of or current treatment for hypertension, coronary heart disease; or angina pectoris; known kidney function issues or disorders; being treated with ACE inhibitors; cancer diagnosis within 5 years of visit; history of chronic disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female male
Study Population: healthy males and females ages 18-64
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-07-13 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Arginine levels in plasma | 0-180 minutes
  Measured blood plasma arginine levels at various time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research, Raritan, New Jersey, United States